CLINICAL TRIAL: NCT03091686
Title: Sedentary Behaviour and Diabetes Information as a Source of Motivation to Reduce Daily Sitting Time in Adult Office Workers: A Pilot Randomized Controlled Trial
Brief Title: The Health Action Process Approach and Movement Patterns in Adult Office Workers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Dr. Harry Prapavessis, Professor, Western University, Canada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HAPA and Sedentary Behaviour
Record Dates: First submitted 2017-03-16; First posted 2017-03-27 (Actual); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Sedentary Lifestyle
Keywords: Sedentary Behaviour; Health Behaviour Change; Health Action Process Approach; Intervention; Prolonged Sitting; Light Intensity Physical Activity; Motivational Factors; Intentions; Diabetes; Self-Efficacy; Risk Perception; Outcome Expectancies
MeSH Terms: conditions — Sedentary Behavior; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental Group (HAPA SB) (Experimental): Experimental (same outcome questionnaire but with informational slideshow focusing on sedentary behaviour and diabetes risk)
  HAPA SB Intervention Slideshow
  Interventions: Behavioral: HAPA SB Intervention Slideshow
- Attention-Control Group (HAPA MVPA) (Active Comparator): Attention-Control (same outcome questionnaire but with slideshow focusing on benefits of moderate-vigorous physical activity)
  HAPA MVPA Intervention Slideshow
  Interventions: Behavioral: HAPA MVPA Attention-Control Slideshow
- Control Group (No Intervention): Control (outcome questionnaire without any slideshow)
  Participants randomly assigned to the control group will receive no information or intervention of any kind and will only be asked to complete the outcome questionnaire.

INTERVENTIONS:
Behavioral: HAPA SB Intervention Slideshow — In the experimental condition, participants will receive sedentary behaviour and diabetes information in the form of a slide show that will be viewed online. The intervention aims to address all components of the Health Action Process Approach. For the experimental group, the intervention material will target risk perceptions (RP) related to sitting by presenting evidence supported by research on sedentary behaviour and diabetes risk; outcome expectancies (OE) by presenting research on the effectiveness of breaking up sedentary time for improving blood sugar and insulin levels; and self-efficacy (SE) by providing strategies on how to reduce and break up sitting time.
  Arms: Experimental Group (HAPA SB)
Behavioral: HAPA MVPA Attention-Control Slideshow — In the attention-control, participants will receive information in the form of a slide show that will be viewed online. The intervention aims to address all components of the Health Action Process Approach. The attention-control slide show will take the same approach as the Experimental group slideshow but the slides will be geared towards meeting moderate-vigorous physical activity guidelines.
  Arms: Attention-Control Group (HAPA MVPA)

SUMMARY:
Societal changes have resulted in reduced demands to be active and increased daily time spent sitting. Excessive sitting has been shown to be a health hazard. The purpose of this study is to examine whether sedentary behaviour and diabetes information grounded in the Health Action Process Approach is a meaningful source of motivation to reduce daily sitting time among adult office workers. The intervention will target risk perceptions related to sitting by presenting research on prolonged sitting and diabetes risk, the effectiveness of breaking up prolonged sitting, and provide strategies to break up sitting. It is expected that participants who receive this information will report greater motivation and intentions to reduce both work and leisure sitting time.

DETAILED DESCRIPTION:
Using a Health Action Process Approach framework, the purpose of this study is to examine whether sedentary behaviour and diabetes information is a meaningful source of motivation to reduce daily sitting time among preintending adult office workers. Specifically, to examine the effectiveness of an intervention guided by HAPA to influence participants' pre-intentional motivational constructs (i.e., sedentary-derived risk perceptions [RP], outcome expectancies [OE], self-efficacy [SE]) and intentions (GI) for reducing both occupational and leisure-time sedentary behaviour.

Sedentary office-workers who had given little thought to how much they sit were targeted to discriminate preintenders from intenders. Research has demonstrated the benefits of matching self-help manuals and other motivational materials to a person's stage of readiness or change (e.g., Graham, Prapavessis, & Cameron, 2006; Pope, Pelletier, & Guertin, 2017)

This is a pilot randomized controlled trial with outcome variables being assessed immediately post-intervention. If successful, participants in the Experimental Group (sedentary intervention group) will report higher outcome expectancies (OE) regarding reducing sitting time, higher risk perceptions (RP) regarding SB and diabetes risk, higher self-efficacy (SE) to reduce both occupational and leisure-time SB, and greater intentions (GI) to reduce both occupational and leisure-time SB at post-intervention, compared to participants in either the Attention-control Group or Control Group. In addition, it is hypothesized that participants in the Attention-control Group, those who received information about the benefits of physical activity, will also show slightly greater scores on pre-intentional motivational factors (i.e., OE, RP, and SE) and behavioural intentions (GI) those those in the Control Group based on the reminder that moderate-vigorous physical activity is important (which implies that sitting should be minimized). Participants in the Control Group are not expected to report any changes in sitting-related motivational factors post-intervention.

This is a pilot randomized controlled trial (RCT) with outcome variables being assessed immediately post-intervention. Participants will be full-time adult, office workers primarily recruited from large businesses and office spaces. Potential participants (estimated enrollment: 252) will be recruited by Andrew Rollo, Co-Investigator, and Harry Prapavessis, Principal Investigator, for this study. Relevant contacts (i.e., Head of Human Resources, President, Chief Executive Officer, Office Manager) at potential businesses of interest will be contacted via email. The email will include the letter of information (LOI) and recruitment poster. If the individual accepts the invitation to participate and informs the researchers that he/she is willing to facilitate and aid with the recruitment process, a face-to-face meeting will be arranged. During this meeting, full and complete study details (i.e., purpose, design, methods and procedure) will be made clear to the ONE individual (i.e., Head of Human Resources, President, CEO, Office Manager). The individual will then be asked to email all full-time employees in the respective office/business and offer them the opportunity to participate. In this recruitment email, brief study details, a recruitment poster and a link to an online survey (i.e., including the Letter of Information, Informed Consent, and online questionnaire) using the SurveyMonkey website will be provided to all employees. Adult office-workers who choose to take part in this study will be asked to complete an online questionnaire using SurveyMonkey. Participants will be assured that participation in this study is voluntary, that they are free to discontinue and withdraw from the study at any time, and that they may choose to skip any questions that they do not wish to answer without any effect on their employment status/work conditions. In other words, refusing to participate, refusing to answer any questions or withdrawing from the study will not impact their employment beyond potentially not receiving benefits associated with study participation. After viewing the Letter of Information and indicating that they consent to participate in the study (by clicking "I agree" on the survey), participants will be asked to complete a brief demographics questionnaire. All participants will then be randomized to one of three groups: Control (outcome questionnaire without any slides), Attention-Control (same outcome questionnaire but with slides focusing on benefits of moderate-vigorous physical activity), or Experimental (same outcome questionnaire but with slides focusing on sedentary behaviour and diabetes risk). Depending on group assignment, participation should take between 30 minutes and 45 minutes total. In the attention-control and experimental condition, participants will receive information in the form of a slide show that will be viewed online. The intervention aims to address all components of the Health Action Process Approach. For the experimental group, the intervention material will target risk perceptions (RP) related to sitting by presenting evidence supported by research on sedentary behaviour and diabetes risk; outcome expectancies (OE) by presenting research on the effectiveness of breaking up sedentary time for improving blood sugar and insulin levels; and self-efficacy (SE) by providing strategies on how to reduce and break up sitting time. The attention-control slide show will take the same approach but the slides will be geared towards meeting moderate-vigorous physical activity guidelines. Participants randomly assigned to the control group will receive no information or intervention of any kind and will only be asked to complete the outcome questionnaire. Regardless of group assignment, all participants will complete the same measures post-intervention (i.e., questionnaire measuring sedentary-related pre-intentional motivational constructs [RP, OE, SE] and intentions [GI]). However, participants in the attention-control and experimental group will FIRST receive information in the form of a slide show that will be delivered online. The first question assesses outcome expectancies (OE) with respect to reducing daily sitting time; the second question assesses risk perceptions (RP) related to sitting time and diabetes risk; questions 3-12 assess self-efficacy (SE) related to reducing sedentary behaviour; and questions 13-22 assess intentions (GI) related to reducing sedentary behaviour. The post-intervention outcome questionnaire will be administered online via SurveyMonkey immediately following intervention delivery (with the exception of control group who will solely complete the questionnaire). All responses are completely confidential.

Only participants who responded 'somewhat' or below in response to the baseline screening question, which asked whether they had given any thought to how much time they spent sitting, were used in the main analyses (n = 96) to test the major hypotheses generated for the present study.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible to participate, participants must be between 18 and 64 years of age, be a full-time worker/employee in an office setting, be able to read and write in English, and have access to a computer with Internet.

Exclusion Criteria:

* Individuals who are not between 18-64 years of age, do not read or write in English, are not full-time workers/employees in office settings, and do not have access to a computer with Internet are not eligible to participate in this study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 218 (Actual)
Dates: Start 2017-08-17 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Participants' intentions to reduce leisure sitting time | Immediately Post-intervention
  Health Action Process Approach sedentary-derived Goal Intention (GIL) 15-items; 5-point scale Five Sub-scale scores (3-items each); GIL1- Intentions to reduce sitting time outside of work; GIL2 - Intentions to increase the number of breaks from sitting outside of work; GIL3 - Intentions to increase the length of breaks from sitting outside of work; GIL4 - Intentions to increase standing time outside of work; GIL5 - Intentions to increase light movement time outside of work
Participants' intentions to reduce occupational sitting time | Immediately Post-intervention
  Health Action Process Approach sedentary-derived Goal Intention (GIO) 15-items; 5-point scale Five Sub-scale scores (3-items each); GIO1- Intentions to reduce sitting time at work; GIO2 - Intentions to increase the number of breaks from sitting at work; GIO3 - Intentions to increase the length of breaks from sitting at work; GIO4 - Intentions to increase standing time at work; GIO5 - Intentions to increase light movement time at work

SECONDARY OUTCOMES:
Participants expectations regarding reducing daily sitting time and improved health outcomes | Immediately Post-intervention
  Health Action Process Approach sedentary-derived pre-intentional motivational construct - Outcome Expectancies (OE) 4-items; 5-point scale
Participants perceptions regarding sitting time and diabetes risk | Immediately Post-intervention
  Health Action Process Approach sedentary-derived pre-intentional motivational construct - Risk Perceptions (RP) 4-items; 5-point scale
Participants confidence to reduce leisure sitting time | Immediately Post-intervention
  Health Action Process Approach sedentary-derived pre-intentional motivational construct - Self-Efficacy (SEL) 55-items; 11-point scale Five Sub-scale scores; SEL1 (12-items) - Confidence to reduce sitting time outside of work; SEL2 (10-items) - Confidence to increase the number of breaks from sitting outside of work; SEL3 (9-items) - Confidence to increase the length of breaks from sitting outside of work; SEL4 (12-items) - Confidence to increase standing time outside of work; SEL5 (12-items) - Confidence to increase light movement time outside of work
Participants confidence to reduce occupational sitting time | Immediately Post-intervention
  Health Action Process Approach sedentary-derived pre-intentional motivational construct - Self-Efficacy (SEO) 55-items; 11-point scale Five Sub-scale scores; SEO1 (12-items) - Confidence to reduce sitting time at work; SEO2 (10-items) - Confidence to increase the number of breaks from sitting at work; SEO3 (9-items) - Confidence to increase the length of breaks from sitting at work; SEO4 (12-items) - Confidence to increase standing time at work; SEO5 (12-items) - Confidence to increase light movement time at work

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Western Ontario, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No